CLINICAL TRIAL: NCT04116983
Title: Effectiveness of an Image Analysing Algorithm (DERM) to Diagnose Non-melanoma Skin Cancer (NMSC) and Benign Skin Lesions Compared to Gold Standard Clinical and Histological Diagnosis
Brief Title: DERM NMSC Validation Study
Status: Completed | Type: Observational
Sponsor: Skin Analytics Limited (Industry)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: DERM-003
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Recruited participants will be attending a dermatology clinic with at least one skin lesion where there is a suspicion of skin cancer. All suspicious lesions suitable for photographing will be photographed six times in a single visit. A macro and dermoscopic image of each lesion will be captured by three different mobile phones: an iPhone, a Samsung and a Nokia smart phone, without (macro image) or with (dermoscopic image) a Dermlite DL1 lens attached. Dermoscopic images of healthy skin will also be captured by each camera. Images of the lesions will be analysed by DERM. The DERM results for lesions biopsied will be compared to the biopsy result; the DERM results for lesions not biopsied will be compared to the clinical assessment.
  Interventions: Device: Deep Ensemble for the Recognition of Malignancy (DERM)

INTERVENTIONS:
Device: Deep Ensemble for the Recognition of Malignancy (DERM) — An AI-based diagnosis support tool

SUMMARY:
This study aims to establish the effectiveness of an Artificial Intelligence (AI) algorithm (DERM) to determine the presence of Basal Cell Carcinoma (BCC) and Squamous Cell Carcinoma (SCC) and frequently observed benign conditions, when used to analyse images of skin lesions taken by commonly available smart phone cameras.

DETAILED DESCRIPTION:
DERM, an Artificial Intelligence (AI)-based diagnosis support tool, has been shown to be able to accurately identify Non-melanoma skin cancers (NMSC) and other conditions from historical images of suspicious skin lesions (moles). This study aims to establish how well DERM determines the presence of these conditions in images of skin lesions collected in a clinical setting.

Suspicious skin lesions that are due to be assessed by a dermatologist and a patch of healthy skin will be photographed using three commonly available smart phone cameras with a specific lens attachment. The images will be analysed by DERM, and the results compared to the clinician's diagnosis (all lesions) and histologically-conformed diagnosis (any lesion that is biopsied).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study,
* Male or Female, aged 18 years or above,
* Have at least suspicious skin lesion which is suitable for photographing (<15mm, not located on an anatomical site inappropriate to photograph (genitalia, hair-bearing areas, under nails), not previously biopsied, not located in an area of visible scarring or tattooing),
* In the Investigator's opinion, able and willing to comply with all study requirements.

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending a dermatology clinic with at least 1 suspicious skin lesion
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
AUROC of DERM performance when analysing images of biopsied lesions | Study completion
  Area Under the Receiver Operating Characteristic Curve (AUROC) of the DERM result of biopsied lesions, using histopathological-confirmed diagnosis as gold standard

SECONDARY OUTCOMES:
AUROC of DERM performance when analysing images of non-biopsied lesions | Study completion: on average 2 days
  Area Under the Receiver Operating Characteristic Curve (AUROC) of the DERM result of biopsied lesions, using clinical diagnosis as gold standard
The sensitivity of DERM when used to assess biopsied lesions | Study completion: on average 2 days
  The sensitivity of DERM when used to assess biopsied lesions
The specificity of DERM when used to assess biopsied lesions | Study completion: on average 2 days
  The specificity of DERM when used to assess biopsied lesions
The false positive rate of DERM when used to assess biopsied lesions | Study completion: on average 2 days
  The false positive rate of DERM when used to assess biopsied lesions
The false negative rate of DERM when used to assess biopsied lesions | Study completion: on average 2 days
  The false negative rate of DERM when used to assess biopsied lesions
The positive predictive value of DERM when used to assess biopsied lesions | Study completion: on average 2 days
  The positive predictive value of DERM when used to assess biopsied lesions
The negative predictive value of DERM when used to assess biopsied lesions | Study completion: on average 2 days
  The negative predictive value of DERM when used to assess biopsied lesions
The sensitivity of DERM when used to assess non-biopsied lesions | Study completion: on average 2 days
  The sensitivity of DERM when used to assess non-biopsied lesions
The specificity of DERM when used to assess non-biopsied lesions | Study completion: on average 2 days
  The specificity of DERM when used to assess non-biopsied lesions
The false positive rate of DERM when used to assess non-biopsied lesions | Study completion: on average 2 days
  The false positive rate of DERM when used to assess non-biopsied lesions
The false negative rate of DERM when used to assess non-biopsied lesions | Study completion: on average 2 days
  The false negative rate of DERM when used to assess non-biopsied lesions
The positive predictive value of DERM when used to assess non-biopsied lesions | Study completion: on average 2 days
  The positive predictive value of DERM when used to assess non-biopsied lesions
The negative predictive value of DERM when used to assess non-biopsied lesions | Study completion: on average 2 days
  The negative predictive value of DERM when used to assess non-biopsied lesions
Concordance of clinician assessment with histologically confirmed diagnosis | Study completion: on average 2 days
  Concordance of clinician assessment with histologically confirmed diagnosis
The concordance of DERM result generated using images from each camera | Study completion: on average 2 days
  The concordance of DERM result generated using images from each camera
The proportion of skin lesions with 3 images that can be analysed by DERM; | Study completion: on average 2 days
  The proportion of skin lesions with 3 images that can be analysed by DERM;
The proportion of skin lesions with at least 1 readable image that can be analysed by DERM | Study completion: on average 2 days
  The proportion of skin lesions with at least 1 readable image that can be analysed by DERM

OTHER OUTCOMES:
Impact of patient characteristics on the DERM and clinician assessment | Study completion: on average 2 days
  The impact of patient characteristics (such as sex, age, location of lesion, total body lesion count, Fitzpatrick skin type, past medical history of skin cancer) on the diagnostic accuracy of DERM and clinician assessment;
Impact of lesion characteristics on the DERM and clinician assessment | Study completion: on average 2 days
  The impact of lesions characteristic (such as growth over last 6 months, stage and sub-type) on the diagnostic accuracy of DERM and clinician assessment
The impact of image variables on the diagnostic accuracy of DERM assessment | Study completion: on average 2 days
  The impact of image variables (such as macro and dermoscopic images) on the diagnostic accuracy of DERM assessment
DERM performance (AUROC) when macro images are used both to train the algorithm and as test images | Study completion: on average 2 days
  Exploration of whether macro images can be used as part of DERM's assessment

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Free London NHS Foundation Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Poole General Hospital, Poole

IPD SHARING:
Plan to Share IPD: Undecided
Research to improve or test the performance of DERM only allowed in consent